CLINICAL TRIAL: NCT02996968
Title: Is Self-discontinuation of a Transurethral Catheter Following Pelvic Reconstructive Surgery as Effective as Office-based Discontinuation?; A Randomized Controlled Trial
Brief Title: Self-discontinuation of a Transurethral Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-075
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-removal group (Experimental): The patients randomized to the self-removal group will be provided with a diagrammatic handout and will be instructed to remove their indwelling urinary catheter at home on the morning of Postoperative day 7.
  Interventions: Procedure: Self-removal
- Office-removal group (No Intervention): The patients randomized to the office-removal group will visit the office for a repeat voiding trial on postoperative day 6-8 (postoperative day 7 will be encouraged). At this visit, the patients will undergo a backfill voiding trial.

INTERVENTIONS:
Procedure: Self-removal — Self-discontinuation of a transurethral catheter
  Arms: Self-removal group

SUMMARY:
This study is to determine if self-discontinuation of transurethral foley catheters in patients diagnosed with postoperative urinary retention (POUR), which is defined as the continued need for catheterization, following impatient pelvic organ prolapse surgery is non-inferior to office-discontinuation.

DETAILED DESCRIPTION:
Postoperative urinary retention (POUR) is a common issue following urogynecologic surgery, with incidence rates of 1.4-43%. The wide range of incidence is due to the lack of a standardized definition of POUR. Generally speaking, POUR can be characterized by any impairment in bladder emptying following surgery. While the gold standard for assessing voiding function remains measurement of a postvoid residual (PVR), there are many voiding trial (VT) methods being used across institutions.

Historically, the most widely accepted postoperative VT for the assessment of voiding function was the backfill method. An alternative assessment of voiding function is the spontaneous VT, where the indwelling catheter is removed and a patient is asked to void spontaneously when a patient has the urge. It is controversial which of these methods are superior, and studies are conflicted. Nevertheless, both of these methods were studied in a clinical setting, and we lack information on self-discontinuation efficacy at home.

Managing an indwelling urinary catheter and returning to the outpatient clinic only a week after discharge from the hospital can be overwhelming for patients and their involved caregivers. Given the low incidence of POUR at one-week postoperative and patient dissatisfaction with urinary catheter management, home self-removal of indwelling urinary catheters is an important topic of investigation.

We are trying to compare the incidence of POUR between self-discontinuation and office-discontinuation of urinary catheters. The results of this study could impact on the decision regarding catheter use following inpatient pelvic organ prolapse surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing vaginal vault suspension or robot-assisted laparoscopic sacrocolpopexy by a physician at Cincinnati Urogynecology Associates, TriHealth Inc.for the treatment of pelvic organ prolapse
* Failed voiding trial prior to discharge
* Concomitant procedures such as hysterectomy, suburethral sling, anterior or posterior colporrhaphy, bilateral salpingectomy or salpingooophorectomy

Exclusion Criteria:

* physical or mental impairment that would affect the subject's ability to self-remove indwelling urinary catheter, including patient's with Multiple Sclerosis, Dementia, Parkinsonism, or those who have impaired mobility or are wheelchair bound
* Bladder injury, fistula repair or other need for prolonged catheterization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shatkin-Margolis A, Yook E, Hill AM, Crisp CC, Yeung J, Kleeman S, Pauls RN. Self-Removal of a Urinary Catheter After Urogynecologic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2019 Nov;134(5):1027-1036. doi: 10.1097/AOG.0000000000003531. PMID 31599827

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-discontinuation Group: The patients randomized to the self-discontinuation group will be provided with a diagrammatic handout and will be instructed to remove their indwelling urinary catheter at home on the morning of Postoperative day 7.
- Office-discontinuation Group: The patients randomized to the office-discontinuation group will visit the office for a repeat voiding trial on postoperative day 6-8 (postoperative day 7 will be encouraged). At this visit, the patients will undergo a backfill voiding trial.
Period: Overall Study
Arm/Group | Self-discontinuation Group | Office-discontinuation Group
Started | 79 | 79
Completed | 78 | 79
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Office-discontinuation Group: The patients randomized to the discontinuation group will visit the office for a repeat voiding trial on postoperative day 6-8 (postoperative day 7 will be encouraged). At this visit, the patients will undergo a backfill voiding trial.
- Total: Total of all reporting groups
Arm/Group | Self-discontinuation Group | Office-discontinuation Group | Total
Number analyzed (Participants) | 78 | 79 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.0) | 60.2 (12.3) | 60.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 79 | 157
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75 | 75 | 150
  Black/African American | 3 | 3 | 6
  Hispanic | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 78 | 79 | 157

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Urinary Retention
Description: Number of Participants with postoperative urinary retention (POUR) following pelvic reconstructive surgery for pelvic organ prolapse.
  Pour at 1-week was defined as continued catheterization on POD 6-8
Time Frame: postoperative day 6-8
Measure: Count of Participants; unit: Participants
Arm/Group | Self-discontinuation Group | Office-discontinuation Group
Number analyzed (Participants) | 78 | 79
Participants | 11 | 11
Statistical Analysis 1: Comparison: Self-discontinuation Group vs Office-discontinuation Group; Test type: Non-Inferiority — Non-inferiority was declared if the POUR rate at 1-week with self-discontinuation was no worse than the POUR rate at 1-week with office-discontinuation, by a pre-specified margin of 15%. A sample size was calculated to be 74 patients in each arm based on the following: * The estimated POUR requiring indwelling urinary catheter at 1-week postoperative is 16% * The non-inferiority margin was set at 15%. * The power was set at 80%; p = 0.5, Two proportions Z-test — 2-sample test for equality of proportions with continuity correction; Proportion Difference = 0.002, 95% CI 1-sided [upper limit 0.095]

ADVERSE EVENTS:
Time Frame: 6 weeks postoperative
Arm/Group | Self-discontinuation Group | Office-discontinuation Group
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/79
Other Adverse Events (participants affected / at risk) | 0/78 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT02996968/Prot_SAP_000.pdf